CLINICAL TRIAL: NCT02829918
Title: A Phase II Investigator Sponsored Study of Nivolumab in Patients With Advanced Refractory Biliary Tract Cancers
Brief Title: Study of Nivolumab in Patients With Advanced Refractory Biliary Tract Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18684
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Biliary Tract Cancer; Biliary Tract Neoplasms
Keywords: advanced biliary tract cancer; refractory biliary tract cancer; digestive diseases; immunotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms; Digestive System Diseases | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nivolumab Treatment (Experimental): This is a single arm study with two stage design using nivolumab in advanced biliary tract cancer (BTC), for participants who have failed or are intolerant to at least one line of therapy and no more than 2 lines of therapy. In the first stage, 18 participants will be accrued. If there is at least one response (or several participants with stable disease based on the study team's discretion), an additional 34 patients will be accrued for a total of 52 patients.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Participants will receive nivolumab at a dose of 240 mg intravenously (IV) every 2 weeks (Q 2W) for 16 weeks (16W) and then 480 every 4 weeks (Q4W) from 17 weeks to end of study.
  Other Names: OPDIVO

SUMMARY:
This research study is designed to see if a drug called Nivolumab is effective in treating patients with advanced refractory biliary tract cancers. Nivolumab has been approved by the U.S. Food and Drug Administration (FDA) for treatment of certain types of cancer but is not approved by the FDA for treatment of your type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically documented carcinoma primary to the intra- or extra-hepatic biliary system or gall bladder with clinical and/or radiologic evidence of unresectable, locally advanced or metastatic disease. Patients with ampullary carcinoma are not eligible.
* Must have failed or are intolerant to one line of systemic treatment but no more than 2 prior lines of systemic chemotherapy for advanced BTC. Patients who received adjuvant chemotherapy and had evidence of disease recurrence within 6 months of completion of the adjuvant treatment are also eligible. If the patient received adjuvant treatment and had disease recurrence after 6 months, patients will only be eligible after failing or having intolerance to one line of systemic chemotherapy used to treat the disease recurrence.
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status Assessment of 0 or 1.
* Must have radiographic measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Life expectancy of at least 12 weeks (3 months).
* For patients who have received prior radiation, cryotherapy, radiofrequency ablation, therasphere, ethanol injection, transarterial chemoembolization (TACE) or photodynamic therapy, the following criteria must be met: 28 days have elapsed since that therapy; Lesions that have not been treated with local therapy must be present and measureable.
* Must be able to understand and be willing to sign the written informed consent form. Must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other study requirements.
* All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF) except for alopecia.
* Adequate bone marrow, liver and liver function.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity of 25 IU/L or equivalent units of HCG) performed within24 hours prior to the start of nivolumab Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Men and women of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 3 months after the last dose of study drug.
* Patients with history of hepatitis B and hepatitis C will be eligible but patients with hepatitis B must be started on antiviral therapy prior to beginning study therapy.
* Availability of archival tumor tissue for biomarkers analysis (FFPE block or cell block will be required).

Exclusion Criteria:

* Active central nervous system (CNS). If CNS metastases are treated and potential participants are at neurologic baseline for at least 2 weeks prior to enrollment, they will be eligible but will need a Brain MRI prior to enrollment. Must be off corticosteroids or on a dose of less than 10 mg per day.
* Active, known or suspected autoimmune disease. Potential participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
* Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Known history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
* Child Pugh B or C disease.
* History of severe hypersensitivity reactions to other monoclonal antibodies.
* History of allergy or intolerance to study drug components or Polysorbate-80-containing Infusions.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
* Unresolved toxicity higher than CTCAE grade1 attributed to any prior therapy/procedure excluding alopecia.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity of 25 IU/L or equivalent units of HCG) performed within 24 hours prior to the start of nivolumab and a negative results must be documented before start of treatment.
* Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study.
* Excluded Therapies and Medications for Cancer: 1) Anticancer chemotherapy during the study or within 4 weeks of study enrollment. Must have recovered from the toxic effects of the previous anti-cancer chemotherapy (with the exception of alopecia). Anti-cancer therapy is defined as any agent or combination of agents with clinically proven anti-tumor activity administered by any route with the purpose of affecting the malignancy, either directly or indirectly, including palliative and therapeutic endpoints. 2) Hormonal therapy during the study or within 2 weeks of first study enrollment. 3) Radiotherapy to target lesions during study or within 2 weeks of enrollment. 4) An irradiated lesion is considered evaluable only if it has shown enlargement since the completion of last radiation. 5) Bone marrow transplant or stem cell rescue. 6) Investigational drug therapy outside of this trial during or within 4 weeks of first study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - City of Hope Cancer Center, Duarte, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia

REFERENCES:
- [Derived] Kim RD, Chung V, Alese OB, El-Rayes BF, Li D, Al-Toubah TE, Schell MJ, Zhou JM, Mahipal A, Kim BH, Kim DW. A Phase 2 Multi-institutional Study of Nivolumab for Patients With Advanced Refractory Biliary Tract Cancer. JAMA Oncol. 2020 Jun 1;6(6):888-894. doi: 10.1001/jamaoncol.2020.0930. PMID 32352498
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center, City of Hope Cancer Center and Winship Cancer Center October 2016 through January 2019.
Groups:
- Nivolumab Treatment: This is a single arm study with two stage design using nivolumab in advanced biliary tract cancer (BTC), for participants who have failed or are intolerant to at least one line of therapy and no more than 2 lines of therapy. In the first stage, 18 participants will be accrued. If there is at least one response (or several participants with stable disease based on the study team's discretion), an additional 34 patients will be accrued for a total of 52 patients.
  Nivolumab: Participants will receive nivolumab at a dose of 240 mg intravenously (IV) every 2 weeks (Q 2W) for 16 weeks (16W) and then 480 mg every 4 weeks (Q4W) from 17 weeks to end of study.
Period: Overall Study
Arm/Group | Nivolumab Treatment
Started | 54
Completed | 46
Not Completed | 8
Not completed — Death | 2
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1
Not completed — Progression | 1

BASELINE CHARACTERISTICS:
Population: 54 participants at baseline, 46 participants were evaluable for outcome measures
Groups:
- Nivolumab Treatment: This is a single arm study with two stage design using nivolumab in advanced biliary tract cancer (BTC), for participants who have failed or are intolerant to at least one line of therapy and no more than 2 lines of therapy. In the first stage, 18 participants will be accrued. If there is at least one response (or several participants with stable disease based on the study team's discretion), an additional 34 patients will be accrued for a total of 52 patients.
  Nivolumab: Participants will receive nivolumab at a dose of 240 mg intravenously (IV) every 2 weeks (Q 2W) for 16 weeks (16W) and then 480 mg Q4W from 17 weeks to end of study.
Arm/Group | Nivolumab Treatment
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 42
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) After 4 Cycles of Treatment
Description: Response in participants with advanced biliary tract cancers receiving nivolumab as a single agent. ORR is defined as complete responses (CR) plus partial responses (PR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Time Frame: 16 weeks
Population: 46 participants were evaluable for response
Measure: Number; unit: percent
Arm/Group | Nivolumab Treatment
Number analyzed (Participants) | 46
percent | 22

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from enrollment to the date of death.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Treatment
Number analyzed (Participants) | 46
months | 8.9 [5.2 to 17]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from first treatment to the date of the first documented tumor progression as determined by the investigator (per RECIST 1.1), or death due to any cause.
Time Frame: Up to 36 months
Population: 46 participants evaluable
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Treatment
Number analyzed (Participants) | 46
months | 3.68 [2.30 to 5.69]

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected from initiation of study drug to a minimum of 30 days from end of treatment. All Serious Adverse Events collected from on treatment date to within 100 days of discontinuation of dosing or until patient begins another anti-cancer therapy, up to 28 months.
Groups:
- Nivolumab Treatment: All participants receiving at least one dose of Nivolumab per protocol.
Arm/Group | Nivolumab Treatment
All-Cause Mortality (participants affected / at risk) | 2/54
Serious Adverse Events (participants affected / at risk) | 32/54
Other Adverse Events (participants affected / at risk) | 52/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab Treatment (N=54)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Death NOS (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 2 (3)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Stroke (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab Treatment (N=54)
Infusion related reaction (General disorders) | 4 (5)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 10 (12)
Weight loss (Investigations) | 18 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (13)
Anemia (Blood and lymphatic system disorders) | 10 (13)
Abdominal pain (Gastrointestinal disorders) | 25 (35)
Edema limbs (General disorders) | 5 (5)
Fatigue (General disorders) | 21 (24)
Alkaline phosphatase increased (Investigations) | 9 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Non-cardiac chest pain (General disorders) | 6 (6)
Lymphocyte count decreased (Investigations) | 9 (14)
Headache (Nervous system disorders) | 4 (4)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 (7)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 12 (14)
Flatulence (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 9 (14)
Hyponatremia (Metabolism and nutrition disorders) | 8 (16)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Blood and lymphatic system disorders -Other (Blood and lymphatic system disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 2 (3)
Skin infection (Infections and infestations) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Ventricular arrhthmia (Cardiac disorders) | 1 (1)
Pain (General disorders) | 3 (3) — Joint Pain
Creatinine increased (Investigations) | 5 (5)
Platelet count decreased (Investigations) | 3 (3)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 9 (14)
Sepsis (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 5 (5)
Blood bilirubin increased (Investigations) | 7 (12)
Hypokalemia (Metabolism and nutrition disorders) | 4 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (5)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (4)
Eye disorders - Other (Eye disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 8 (9)
Nausea (Gastrointestinal disorders) | 10 (15)
Vomiting (Gastrointestinal disorders) | 13 (20)
White blood cell decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Hypertension (Vascular disorders) | 8 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Hypotension (Vascular disorders) | 6 (7)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 4 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Investigations -Other (Investigations) | 1 (1) — Elevated creatinine
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (9)
Anorexia (Metabolism and nutrition disorders) | 12 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Allergic reaction (Immune system disorders) | 2 (2)
Hypoalbumenemia (Metabolism and nutrition disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5 (5)
Urinary retention (Renal and urinary disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 4 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Blurred vision (Eye disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (5)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Weight gain (Investigations) | 7 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — Altered mental status
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Papulopustular rash (Infections and infestations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02829918/Prot_SAP_000.pdf